CLINICAL TRIAL: NCT06615141
Title: Immersive Versus Non-immersive Virtual Reality in Enhancing Upper Limb Functions Among Individuals With Subacute Stage Hemiplegia - A Randomized Controlled Trial
Brief Title: Immersive v/s Non-immersive Virtual Reality in Enhancing Upper Limb Functions Among Individuals With Subacute Stage Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Athira George, Principal Investigator, Gulf Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-75-FEB-2024
Record Dates: First submitted 2024-09-15; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke
Keywords: virtual reality; hemiplegic stroke; Oculus Quest 3; Motor function; Upper limb

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy + Immersive Virtual Reality Therapy (Experimental): 15 minutes of conventional therapy followed by 45 minutes of immersive virtual reality therapy will be administered to this group referred to as Group 1.
  Interventions: Device: Oculus Quest 3
- Conventional Therapy + Non Immersive Virtual Reality Therapy (Experimental): 15 minutes of conventional therapy followed by 45 minutes of non-immersive virtual reality therapy will be administered to this group referred to as Group 2
  Interventions: Device: Neofect Smartboard and Tyromotion Myro

INTERVENTIONS:
Device: Oculus Quest 3 — Oculus quest 3 is a standalone virtual reality headset developed by Meta. It offers precise motion tracking and offers an innovative intervention for stroke rehabilitation, enhancing upper limb motor function throug task - specific exercises.
  Arms: Conventional Therapy + Immersive Virtual Reality Therapy
Device: Neofect Smartboard and Tyromotion Myro — Neofect Smart Board provides non-immersive VR rehabilitation through gamified, task specific exercises to improve upper limb mobility in an interactive way.
  Tyromotion Myro uses non-immersive VR therapy combining sensor-based feedback and interactive games to enhance fine motor skills.
  Arms: Conventional Therapy + Non Immersive Virtual Reality Therapy

SUMMARY:
The goal of this randomized controlled trial is to compare the effectiveness of immersive virtual reality combined with conventional therapy to the effectiveness of non-immersive virtual reality combined with conventional therapy in enhancing upper limb function in subacute hemiplegic stroke patients.

DETAILED DESCRIPTION:
The study is a single blinded randomized controlled trial in which the assessor will be blinded. Male and female participants aged between 28-55 years are included in the study. Participants are selected based on inclusion and exclusion criteria and are later randomly assigned to Group 1 and Group 2.

Group 1 - Conventional therapy and Immersive Virtual Reality Group 2 - Conventional therapy and Non-Immersive Virtual Reality

Primary Outcome measures include the Fugl Meyer Assessment for Upper limb and Graded Wolf Motor Function test for upper limb.

Secondary Outcome measure is the Stroke Specific Quality of Life Scale (SS-QOL) Questionnaire.

Therapy session starts with 15 minutes of stretching and strengthening exercises of the affected arm followed by 45 minutes of Immersive / Non Immersive virtual reality training.

Follow up assessment is done 6 weeks post intervention.

The baseline assessment score and follow up assessment scores will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 28-55 years.
* Diagnosed with hemiplegia due to stroke.
* ≤ Grade 2 on Modified Ashworth scale.
* ≤ Stage 2 on Brunnstrom stages of motor recovery.
* Score of ≥ 35/36 on Cognitive assessment scale for stroke patients (CASP)

Exclusion Criteria:

* Contraindications for VR therapy, such as severe motion sickness or photosensitive epilepsy, impaired spatial awareness.
* Pre-existing neurological conditions such as spinal cord injury, Multiple sclerosis and so affecting upper limb function.

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-01-05 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity (FMA-UE) | From enrollment to the end treatment at 6 weeks
  A valid, reliable, and comprehensive measurement tool with an intra-rater reliability of ICC 0.96 and interrater reliability of ICC 0.98, used to evaluate motor impairment, balance, sensation, and joint function in the upper extremities after stroke.
Graded Wolf Motor function test - The WMFT | From enrollment to the end treatment at 6 weeks
  This test is designed to assess motor function, strength, and coordination in individuals with upper extremity impairments. It is a reliable measure with inter-rater reliability of 0.97 and intra-rater reliability of 0.90.

SECONDARY OUTCOMES:
Stroke Specific Quality of Life Scale (SS-QOL) | From enrollment to the end treatment at 6 weeks
  The SS-QOL scale is widely used for assessing the health-related quality of life in stroke survivors. It has a good test-retest reliability, with ICC ranging from 0.80-0.90. It is a valid and reliable tool for assessing the quality of life in stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Athira George, Master of Physical Therapy, Principal Investigator — Gulf Medical University
Locations (1):
- Thumbay Physical Therapy and Rehabilitation Hospital, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Confidentiality of patient data must be maintained as per consent form.

REFERENCES:
- [Derived] George A, Durairaj SK, Kandakurti PK, Hazari A. Immersive versus non-immersive virtual reality in improving upper limb function among individuals with subacute hemiplegia: a randomized controlled trial. BMC Neurol. 2025 Dec 28. doi: 10.1186/s12883-025-04588-5. Online ahead of print. PMID 41455908